CLINICAL TRIAL: NCT06508970
Title: The Effect of RAM-Based Virtual Reality Glasses Application on Adaptation, Life Satisfaction, and Psychological Well-Being in the Elderly
Brief Title: RAM-Based Virtual Reality Glasses and Adaptation, Satisfaction, Well-Being in the Elderly
Acronym: RAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Gönül GÖKÇAY, Asist. Prof., Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 818295502.903/6
Record Dates: First submitted 2024-07-06; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Nursing; Evidence-Based Nursing
Keywords: Elderly; Roy adaptation model; adaptation difficulty in the elderly; psychological well-being; virtual reality glasses; virtual reality
MeSH Terms: conditions — Psychological Well-Being | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Intervention Model Description: RAM-based virtual reality glasses were applied to the experimental group for 4 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were assigned to groups using the "simple randomization method." Participants were not informed about which group they were in. Unique 2-group columns were created with the registration numbers of elderly individuals in nursing homes by using the Random Integer Generator method under the numbers subheading on the Random.org website. The researcher was blind to all conditions until participants started the computer program and the intervention began. Participants were also unaware of whether the group they were assigned to was an experimental or control group. Additionally, researchers who coded and analyzed the data were blinded to randomization and interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): RAM-based virtual reality glasses were applied to the experimental group for 4 weeks.
  Interventions: Behavioral: Experimental RAM-based virtual reality glasses; Other: pre-post test
- Control group (Other): Nursing students will receive their regular semester courses; no additional intervention will be implemented.
  Interventions: Other: pre-post test

INTERVENTIONS:
Behavioral: Experimental RAM-based virtual reality glasses — RAM-based virtual reality glasses were applied to the experimental group for 4 weeks.
  Video contents:
  1. week; 1st sub-dimension (physiological domain)
  2. weeks; 2nd sub-dimension (self-space) Three weeks; 3rd sub-dimension (Role function/function area) week 4; 4th sub-dimension (Independence and interdependence/autonomy)
  Arms: experimental group
Other: pre-post test — Adaptation Difficulty Assessment Scale in the Elderly, Life Satisfaction Scale in the Elderly , and Psychological Well-Being Scale in the Elderly

SUMMARY:
The main purpose of this study is to determine the effect of Roy adaptation model-based virtual reality glasses application on adaptation difficulties, life satisfaction, and psychological well-being in the elderly using a randomized controlled experimental method.

The hypotheses of the study are:

H1: The Roy adaptation model-based virtual reality glasses application has an effect on adaptation difficulties in the elderly.

H2: The Roy adaptation model-based virtual reality glasses application has an effect on life satisfaction in the elderly.

H3: The Roy adaptation model-based virtual reality glasses application has an effect on psychological well-being in the elderly.

DETAILED DESCRIPTION:
In the 21st century, advances in science and technology have led to demographic changes, resulting in an increase in the elderly population. In this process, developments in the field of health such as increased preventive health services and early diagnosis and treatment of diseases played an important role. Aging is a natural process and can be defined as a decrease in an individual's physical and spiritual functions and an increase in external dependency. Adapting the elderly to this period supports psychological well-being by increasing functionality and life satisfaction. The Roy Adaptation Model aims for nurses to meet the needs of individuals to adapt, and this model can also be applied to the elderly. With technological advances, innovations such as virtual reality are used in the field of health and help improve the quality of life of the elderly. In the literature, studies examining the effects of Roy Adaptation Model and virtual reality glasses application on adaptation difficulties, life satisfaction and psychological well-being in the elderly are limited. This study aims to determine the effects of Roy Adaptation Model and virtual reality glasses application on adaptation difficulties, life satisfaction and psychological well-being in the elderly and to lay the foundation for evidence-based research. The thesis is a pre-posttest randomized controlled study with experimental and control groups. In the thesis study, data were collected as pre-post test from the elderly living in nursing homes using the Personal Information Form, Adaptation Difficulty Assessment Scale in the Elderly, Life Satisfaction Scale in the Elderly, and Psychological Well-Being Scale in the Elderly.In the thesis study, the experimental group was shown educational videos and nature videos with VR SHINECON 360 degree virtual reality glasses, based on the Roy adaptation model adaptation areas titles (physiological needs, self-concept area, role function area, interdependence area) twice a week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 60 and over
* Residents of Kocaeli nursing home
* Those who score 25 and above in the Standardized Mini Mental Test

Exclusion Criteria:

* Not wanting to participate in the research voluntarily
* Those who score 24 or below on the Standardized Mini Mental Test

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Adaptation Difficulty Assessment Scale in the Elderly | one months
  It is a 4-point Likert type scale consisting of 24 items, developed and validated by Şişman and Kutlu (2016) according to the Roy Adaptation Model, to determine the adequacy of elderly individuals in adapting to old age. Cronbach Alpha value is 0.93.The individual's compliance level is determined by adding up the total scores from the scale and dividing by the number of items. The lowest possible score is 0 and the highest is 3. It is seen that as the score obtained from the scale increases, the individual's adaptation level to old age decreases.
Life Satisfaction Scale for the Elderly | one months
  It was developed by Altay and Çalmaz in 2022. It has 14 items and 3 subscales that question the participation of elderly individuals in the process related to life satisfaction. Cronbach Alpha value is 0.874. The subscales of the Scale are represented by factors 1, 2 and 3: Self-acceptance (Factor 1), Motivation (Factor 2), Peace of mind (Factor 3). Responses to the items on this 5-point Likert scale are "I strongly disagree" and "I strongly agree". Each item is scored between 1 and 5. The total possible minimum score from the scale is 14, and the highest score that can be obtained is 70. It is known that life satisfaction increases as the score obtained from the scale increases.
Psychological Well-Being Scale in the Elderly | one months
  The scale developed by Gümüş Demir in 2022 consists of fifteen items. In line with the scoring of the scale, no cut-off score has been determined for the level of well-being in the elderly. The Cronbach's alpha internal consistency coefficient of the scale is 0.89. The scale was prepared using a 5-point Likert type response system and the score range varies between 15 and 75. High scores indicate an increase in the level of well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Eda ERSARI ŞEN, Student, Principal Investigator — Kafkas University-Kafkas University Faculty of Health Sciences; Gönül GÖKÇAY, Asist. Prof., Study Director — Bayan.
Locations (1):
- Kafkas University Faculty of Health Sciences, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aydogdu O, Tastan S, Kublay G. The effects of the instrumental reminiscence therapy based on Roy's adaptation model on adaptation, life satisfaction and happiness in older people: A randomized controlled trial. Int J Nurs Pract. 2023 Jun;29(3):e13101. doi: 10.1111/ijn.13101. Epub 2022 Aug 24. PMID 36003030
- [Result] Barsasella D, Liu MF, Malwade S, Galvin CJ, Dhar E, Chang CC, Li YJ, Syed-Abdul S. Effects of Virtual Reality Sessions on the Quality of Life, Happiness, and Functional Fitness among the Older People: A Randomized Controlled Trial from Taiwan. Comput Methods Programs Biomed. 2021 Mar;200:105892. doi: 10.1016/j.cmpb.2020.105892. Epub 2020 Nov 29. PMID 33280934
- [Result] Skjaeret N, Nawaz A, Morat T, Schoene D, Helbostad JL, Vereijken B. Exercise and rehabilitation delivered through exergames in older adults: An integrative review of technologies, safety and efficacy. Int J Med Inform. 2016 Jan;85(1):1-16. doi: 10.1016/j.ijmedinf.2015.10.008. Epub 2015 Oct 28. PMID 26559887